CLINICAL TRIAL: NCT03298074
Title: Apatinib Plus Etoposide Versus Etoposide Alone for Platinum-resistant Recurrent Ovarian Cancer: A Randomized Controlled Trial
Brief Title: Apatinib Plus Etoposide Versus Etoposide Alone for Platinum-resistant Recurrent Ovarian Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Yang Zhijun (Other)
Responsible Party: Sponsor-Investigator, Yang Zhijun, Associate chief physician, Guangxi Medical University
Organization: Guangxi Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HRGX-001
Record Dates: First submitted 2017-09-27; First posted 2017-09-29 (Actual); Last update posted 2017-09-29 (Actual); Status verified 2017-09

CONDITIONS: Ovarian Cancer
Keywords: platinum-resistant; recurrent
MeSH Terms: conditions — Ovarian Neoplasms; Recurrence | interventions — apatinib; Etoposide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Apatinib plus Etoposide (Experimental): Apatinib,500mg,PO.QD, continuous administration Etoposide,100mg, PO.QD，D1-D10, Q3W
  Interventions: Drug: Apatinib; Drug: Etoposide
- Etoposide (Active Comparator): Etoposide,100mg, PO.QD，D1-D10, Q3W
  Interventions: Drug: Etoposide

INTERVENTIONS:
Drug: Apatinib — Apatinib, 500mg,po qd for continuous administration
  Other Names: Aitan
  Arms: Apatinib plus Etoposide
Drug: Etoposide — Etoposide,100mg, PO.QD，D1-D10, Q3W

SUMMARY:
It is a prospective multi-center trial, platinum-resistant ovarian cancer patients will be randomized in two groups, one group will be treated with Apatinib plus Etoposide, the other will be treated with Etoposide alone. It is aimed to see the efficacy and safety of Apatinib plus Etoposide for the platinum-resistant ovarian cancer patients

DETAILED DESCRIPTION:
It is a randomized controlled trial, the aim is to see the efficacy and safety of Apatinib plus Etoposide treating platinum-resistant ovarian cancer. The main primary end point is DCR (disease control rate), the secondary endpoint is Duration of response（DOR），overall survival (OS), time to progression (TTP)，quality of life (QoL, according to EORTC QLQ-C30).The key safety indicators include the patients' vital signs, laboratory indicators, adverse events(AE),serious adverse events.

The data collection duration is from the day ICF assigned to the day(30 days after the end of the last medication).From the day ICF signed to the end of the study, all adverse events were recorded in the CRF. The severity of the adverse events will be evaluated according to the NCI CTCAE 4.0 standard.Each patient will receive a planned visit and specific data at different points will be recorded in the visit.

The patients will be followed up after quitting the trial because of disease progression or intolerance. The following parameters were recorded during follow-up: disease recurrence,metastasis,death time,SAE occurred during the study; survival (available with telephone follow-up, record required).

Adverse events that have not been recovered when the drug is discontinued should be tracked and finalized. All patients should undergo a 30-day follow-up after the last medication to find any new adverse events.

All cases should be recorded carefully and completely, the investigator should be responsible for the authenticity of the center's data.

During the clinical trial, the inspector should send the CRF to the data management unit (in batches), the data administrator will carry out the independent double entry, and carry out the double verification.

The trial as an exploratory test, using a small sample comparison, the test plans to enroll a total of 60 cases.

The statistical analysis plan includes case analysis,demographic data and baseline analysis,efficacy analysis and safety analysis.All statistical tests will be performed on both sides, the difference between the tests was considered statistically significant with a P value less than or equal to 0.05,

ELIGIBILITY:
Inclusion Criteria:

* ECOG PS：0-2 points
* Platinum-resistant recurrent ovarian cancer patients with measurable recurrent focus
* The damage caused by other treatment has been restored (NCI-CTCAE 4.0 Graded ≤ 1 level), Other cytotoxic drugs treatment, radiotherapy or surgery≥ 4 week; EGFR TKI treatment ≥ 2 week
* Baseline routine blood test and biochemical indicators meet the following criteria:

  * Hemoglobin ≥ 90g / L
  * Neutrophil absolute count (ANC) ≥ 1.5 × 109 / L
  * Platelets ≥80 × 109 / L
  * ALT, AST ≤ 2.5 × ULN or 5 × ULN (with liver metastases)
  * Total Serum bilirubin ≤ 1.5 × ULN
  * Serum creatinine≤1.5×ULN or endogenous creatinine clearance ≥ 45ml/min (according to Cockcroft-Gault formula);
* No blood and blood products transfusion in 14 Days
* Expected survival time≥3 month;
* Subjects volunteer to join the study, sign informed consent, cooperate with follow-up.

Exclusion Criteria:

* "biochemical recurrence " ovarian cancer patients
* Patients allergy to apatinib, etoposide and / or its excipients
* Patients with high blood pressure and who can not be reduced to normal range by antihypertensive therapy (systolic blood pressure> 140 mmHg, diastolic blood pressure> 90 mmHg), with grade I coronary heart disease, grade I arrhythmia (including QTc prolongation > 470 ms)
* According to NYHA standard, grade Ⅲ-Ⅳ heart failure, or cardiac color Doppler ultrasound examination shows left ventricular ejection fraction (LVEF) <50%
* Urine protein positive patients
* With a variety of factors that affect oral medication (such as can not swallow, nausea, vomiting, chronic diarrhea and intestinal obstruction, etc.)
* Patients with definite gastrointestinal bleeding tendencies, including the following: localized ulcer lesions, and fecal occult blood (++); 2 months with black stool, hematemesis history
* Patients with coagulation dysfunction (INR> 1.5, APTT> 1.5 ULN), bleeding tendency
* Existing hereditary or acquired bleeding and thrombotic tendencies (such as hemophilia, coagulation disorders, thrombocytopenia, hypersplenism, etc.)
* Long untreated wound or fracture;major surgery or severe traumatic injury in 4 weeks, fracture or ulcer
* Accompanied by abdominal fistula, gastrointestinal perforation or abdominal abscess; active hepatitis B virus or hepatitis C patients
* Active brain metastases, cancer meningitis, spinal cord compression patients, Imaging CT or MRI examination found the brain or pia mater disease,( brain metastases patients who has complete treatment 21 days before and has stable symptoms can be enrolled , but the need for transcranial MRI, CT or intravenous angiography evaluation confirmed as no cerebral hemorrhage symptoms)
* Imaging (CT or MRI) shows tumor lesions from large vessels ≤ 5 mm, or lesions invade the Local large blood vessels
* Lactating women
* Patients with other malignancies in 5 years (except for cured skin basal cell carcinoma and in situ ovarian cancer)
* Patients with a history of psychiatric abuse and who can not quit or have mental disorders
* Patients who participated in other drug clinical trials within 4 weeks
* Patients who received VEGFR inhibitors such as sorafenib and sunitinib treatment
* Patients who received Etoposide treatment
* According to the researcher's judgment, there are serious illnesses that endanger the patient's safety or affect the completion of the study
* Patients that are not suitable for this trial in the investigator's opinions.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — female patient with recurrent ovarian cancer
Enrollment: 60 (Estimated)
Dates: Start 2017-10 (Estimated); Primary Completion 2018-10 (Estimated); Study Completion 2019-04 (Estimated)

PRIMARY OUTCOMES:
Disease Control Rate | through study completion, an average of 1.5 years
  the proportion of patients who had a best response rating of complete response, partial response, or stable disease

SECONDARY OUTCOMES:
Duration of Response | through study completion, an average of 1.5 years
  the time course from the first time tumor assessed as CR or PR to the first time tumor assessed as progressive disease or death
Overall Survival | through study completion, an average of 3 years
  From the beginning of randomization to the cause of death for any reason
Time to Progression | through study completion, an average of 1.5 years
  From randomization to the onset of disease progression or death

CONTACTS AND LOCATIONS:
Overall Officials: Zhijun Yang, Principal Investigator — Affiliated Cancer Hospital & Institute of Guangzhou Medical University

IPD SHARING:
Plan to Share IPD: Undecided